CLINICAL TRIAL: NCT06810089
Title: Examination of Lacrimal Sac and Nasal Mucosa Preparations Taken in Dacryocystorhinostomy Surgery of Patients With Nasolacrimal Duct Obstruction and Comparison of Clinical Groups With Each Other
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Sertac Argun Kivanc, Prof Dr, MD, Uludag University
Other Study IDs: TTU-2023-1352
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-05

CONDITIONS: Dacryocystitis; Dacryocystitis; Chronic; Dacryocystorhinostomy; Epiphora; Nasolacrimal Duct Obstruction; Surfactant; Mucin; Lacrimal Sac Mucosa; Nasal Mucosa
Keywords: dacryocystitis; dacryocystorhinostomy; epiphora; nasolacrimal duct obstruction; staining; mucin; surfactant; immunohistochemical
MeSH Terms: conditions — Dacryocystitis; Bronchiolitis Obliterans Syndrome; Lacrimal Apparatus Diseases; Lacrimal Duct Obstruction; Medullary cystic kidney disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples Without DNA — Nasal mucosa specimen and nasolacrimal sac specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary Nasolacrimal Duct Obstruction without any dacryocystitis history: Immunohistochemical staining scores of nasal mucosa nad nasolacrimal sac mucosa specimens of Primary Nasolacrimal Duct Obstruction without any dacryocystitis history who underwent external dacryocystorhinostomy surgery were compared with other groups. In this group, there were no membranes in the lacrimal sac during the surgery.
- Primary Nasolacrimal Duct Obstruction with dacryocystitis history: In this group patients has had at least one dacryocystitis history. Immunohistochemical staining scores of nasal mucosa nad nasolacrimal sac mucosa specimens of Primary Nasolacrimal Duct Obstruction with dacryocystitis history who underwent external dacryocystorhinostomy surgery were compared with other groups. In this group, there were no membranes in the lacrimal sac during the surgery.
- Traumatic Nasolacrimal Duct Obstruction: In this group, there were patients has traumatic nasolacrimal duct obstruction. Immunohistochemical staining scores of nasal mucosa and nasolacrimal sac mucosa specimens of Secondary Nasolacrimal Duct Obstruction who underwent external dacryocystorhinostomy surgery were compared with other groups. In this group, there were no membranes in the lacrimal sac during the surgery.
- Nasolacrimal Duct Obstruction with Membranes in the Nasolacrimal Sac: In this group, dense membrane was detected in the nasolacrimal sacs during surgery. Patients with and without previous dacryocystitis who were detected to have membranes in their sacs during surgery were evaluated in this group. Immunohistochemical staining scores of nasal mucosa and nasolacrimal sac mucosa specimens of Nasolacrimal Duct Obstruction who underwent external dacryocystorhinostomy surgery were compared with other groups.

SUMMARY:
The goal of this observational study is to investigate etiology and pathogenesis of nasolacrimal duct obstruction and dacryocystitis in different adult clinic groups. The main question it aims to answer is:

Are there differences in terms of staining scores between groups?

There are 4 groups:

Cohort 1: Primary Nasolacrimal Duct Obstruction without any dacryocystitis history Cohort 2: Primary Nasolacrimal Duct Obstruction with dacryocystitis history Cohort 3:Traumatic Nasolacrimal Duct Obstruction Cohort 4:Nasolacrimal Duct Obstruction with Membranes in the Nasolacrimal Sac

DETAILED DESCRIPTION:
One of the most common complaints encountered by patients in the field of eye diseases is epiphora, or watery eyes. The most important cause of watery eyes is nasolacrimal duct obstruction (NLDO), which we frequently encounter in ophthalmology practice. NLDO is usually seen in older ages and in women, but the etiology is not fully known in the primary group. The only treatment for NLDO is surgery. The MOST successful surgical method is external dacryocystorhinostomy (ex-DCR). In this study, the pathology samples routinely taken during ex-DCR surgery from patients who apply to our clinic with NLDO will be re-examined in the Department of Pathology, and the preparations of those who meet the inclusion criteria will be taken and divided into clinical groups. Pathology samples will be examined by staining with hematoxylin & eosin, periodic acid schiff and various immunohistochemical stainings.

The study included adult patients aged 18 years and older who underwent external DCR surgery in our clinic between January 2020 and December 2022 for nasolacrimal duct obstruction and who had lacrimal sac and nasal mucosa samples obtained during surgery. Specimens are investigated prospectively .

It was aimed to examine the preparations taken during surgery of patients who underwent external dacryocystorhinostomy (DCR) surgery due to nasolacrimal duct obstruction (NLDO) by staining them with immunohistochemical staining methods for further research and to compare the clinical groups with each other.

ELIGIBILITY:
Inclusion Criteria:The study included adult patients aged 18 years and older who underwent external DCR surgery in Ophthalmology Department between January 2020 and December 2022 for nasolacrimal duct obstruction and who had lacrimal sac and nasal mucosa samples obtained during surgery.

-

Exclusion Criteria:Patients younger than 18 years of age, and patients in whom lacrimal sac and nasal mucosa were not sampled during surgery were not included in our study. In addition, patients whose outpatient and clinical examination notes were not sufficient for the study and patients who did not attend at least two postoperative follow-up examinations were not included in the study. Patients whose pathology blocks were not accessible in the Department of Pathology and patients with pathology blocks that were not suitable for histopathologic examination due to crush artifact or insufficient tissue in the preliminary examination were not included in our study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to Bursa Uludağ University, School of Medicine, Department of Ophthalmology due to nasolacrimal duct obstruction and underwent external dacryocystorhinostomy surgery and had nasal mucosa and lacrimal sac mucosa samples taken were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Obtaining nasolacrimal sac and nasal mucosa staining scores | 12 months
  Obtaining nasolacrimal sac and nasal mucosa staining scores is the primary outcome measure of this study. Comparison of the staining scores of hematoxylin and eosin, Periodic Acid-Schiff and various immunohistochemical markers will be made between the study groups. It will be investigated whether there is a significant difference between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, School of Medicine, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Provide information about individual participant data may not be accepted by Institutional Review Board